CLINICAL TRIAL: NCT03829787
Title: Attentional Biases, Reward Sensitivity, and Cognitive Control in Adults With Bipolar Disorder and Different Psychiatric Comorbidities: An Eye-Tracking Study
Brief Title: Attentional Biases, Reward Sensitivity, and Cognitive Control in Adults With Bipolar Disorder
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Keming Gao, Director, Mood and Anxiety Clinic, University Hospitals Cleveland Medical Center
Other Study IDs: 09-17-03
Record Dates: First submitted 2018-07-10; First posted 2019-02-04 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Bipolar without Anxiety or Substance Use Disorder: Subjects who are diagnosed with bipolar disorder but do not have any current anxiety or substance use disorders
  Interventions: Device: Eye tracking
- Bipolar disorder with a current anxiety disorder only: Subjects who are diagnosed with bipolar disorder and a current anxiety disorder (generalized anxiety disorder, panic disorder, and/or social phobia) but not a current substance use disorders
  Interventions: Device: Eye tracking
- Bipolar disorder with a current anxiety disorder and a current: Subjects who are diagnosed with bipolar disorder and a current anxiety disorder (generalized anxiety disorder, panic disorder, and/or social phobia) AND a current substance use disorders
  Interventions: Device: Eye tracking
- Bipolar disorder with a current substance use disorder only: Subjects who are diagnosed with bipolar disorder & a substance use disorders but not a current anxiety disorder
  Interventions: Device: Eye tracking
- Healthy Volunteers
  Interventions: Device: Eye tracking

INTERVENTIONS:
Device: Eye tracking — Subjects will be assessed for attentional biases, reward sensitivity, and cognitive control using eye tracking technology

SUMMARY:
The purpose of this study is to use eye-tracking technology to study attentional biases, reward sensitivity, and cognitive control in adult patients with bipolar disorder with or without anxiety and/or substance use disorder comorbidity.

ELIGIBILITY:
1. Inclusion and Exclusion Criteria for Group 1: bipolar disorder without current anxiety or substance use disorder

   1. Inclusion Criteria for Group 1:

   i. Male or female, age 18 or older

   ii. Meets diagnostic criteria for lifetime bipolar I or II disorder according to Diagnostic and Statistical Manual-5 (DSM-5) criteria, as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   iii. Currently in a depressive episode or currently in remission from a mood episode

   iv. Young Mania Rating Scale total score ≤ 8

   v. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   vi. In the opinion of the investigator, has the competency to understand and sign the informed consent

   vii. Subject is compliant with taking psychiatric medication(s) per the investigator's discretion

   b. Exclusion Criteria for Group 1:

   i. Significant structural brain lesion (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Any current psychiatric disorder (other than a current depressive episode) including anxiety disorders, substance use disorders, antisocial personality disorder and borderline personality disorder as assessed by the MINI and clinician assessment.

   iv. Currently pregnant or planning to become pregnant

   v. Tests positive for illegal substances or prescription medications for which they do not have a valid prescription

   vi. Currently taking any steroids, stimulants, or opioid pain killers.

   vii. Meets DSM-5 criteria for any alcohol and/or drug use disorder within the last 6 months, excluding the use of caffeine.Currently experiencing nicotine use disorder or any smoking of cigarettes or use of other nicotine containing products within a week before the eye tracking visit.

   viii. Has had electroconvulsive therapy (ECT) treatment within the last 6 months.
2. Inclusion and Exclusion Criteria for Group 2: Bipolar disorder with a current anxiety disorder (generalized anxiety disorder, panic disorder, and/or social phobia)

   a. Inclusion Criteria for Group 2:

   i. Male or female, age 18 or older

   ii. Meets diagnostic criteria for lifetime bipolar I or II disorder according to DSM-5 criteria, as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   iii. Currently in a depressive episode or currently in remission from a mood episode

   iv. Meets diagnostic criteria for a current anxiety disorder (generalized anxiety disorder, panic disorder, and/or social phobia) as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   v. Hamilton Anxiety Rating Scale total score ≥ 18

   vi. Young Mania Rating Scale total score ≤ 8

   vii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   viii. In the opinion of the investigator, has the competency to understand and sign the informed consent

   ix. Subject is compliant with taking psychiatric medication(s) per the investigator's discretion

   b. Exclusion Criteria for Group 2:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Any co-occurring lifetime or current obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), or attention deficit hyperactivity disorder (ADHD)

   iv. Meets criteria for antisocial personality disorder or borderline personality disorder as assessed by clinician assessment.

   v. Currently pregnant or planning to become pregnant

   vi. Tests positive for illegal substances or prescription medications for which they do not have a valid prescription

   vii. Currently taking any steroids, stimulants, or opioid pain killers.

   viii. Meets DSM-5 criteria for any alcohol and/or drug use disorder within the last 6 months, excluding the use of caffeine

   ix. Currently experiencing nicotine use disorder or any smoking of cigarettes or use of other nicotine containing products within a week before the eye tracking visit.

   x. Has had ECT treatment within the last 6 months.
3. Inclusion and Exclusion Criteria for Group 3: Bipolar disorder with a current anxiety disorder and a current substance use disorder

   a. Inclusion Criteria for Group 3:

   i. Male or female, age 18 or older

   ii. Meets diagnostic criteria for lifetime bipolar I or II disorder according to the DSM-5 criteria, as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   iii. Meets diagnostic criteria for a substance use disorder within the last 3 months

   iv. Meets diagnostic criteria for a current anxiety disorder (generalized anxiety disorder, panic disorder, and/or social phobia) as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   v. Currently in a depressive episode or currently in remission from a mood episode

   vi. Hamilton Anxiety Rating Scale total score ≥ 18

   vii. Young Mania Rating Scale total score ≤ 8

   viii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   ix. In the opinion of the investigator, has the competency to understand and sign the informed consent

   x. Subject is compliant with taking psychiatric medication(s) per the investigator's discretion

   b. Exclusion Criteria for Group 3:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Any co-occurring lifetime or current obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), or attention deficit hyperactivity disorder (ADHD)

   iv. Meets criteria for antisocial personality disorder or borderline personality disorder as assessed by clinician assessment.

   v. Intoxicated or in acute withdrawal state.

   vi. Currently pregnant or planning to become pregnant.

   vii. Currently experiencing nicotine use disorder or any smoking of cigarettes or use of other nicotine containing products within a week before the eye tracking visit.

   viii. Has had ECT treatment within the last 6 months.
4. Inclusion and Exclusion Criteria for Group 4: Bipolar disorder without an anxiety disorder but with a current substance use disorder

   a. Inclusion Criteria for Group 4:

   i. Male or female, age 18 or older

   ii. Meets diagnostic criteria for lifetime bipolar I or II disorder according to the DSM-5 criteria, as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   iii. Meets diagnostic criteria for a substance use disorder within the last 3 months

   iv. Currently in a depressive episode or currently in remission from a mood episode

   v. Young Mania Rating Scale total score ≤ 8

   vi. Hamilton Anxiety Rating Scale total score ≤ 12

   vii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   viii. In the opinion of the investigator, has the competency to understand and sign the informed consent

   ix. Subject is compliant with taking psychiatric medication(s) per the investigator's discretion

   b. Exclusion Criteria for Group 4:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Any co-occurring current anxiety disorder or attention deficit hyperactivity disorder (ADHD)

   iv. Meets criteria for antisocial personality disorder or borderline personality disorder as assessed by clinician assessment.

   v. Intoxicated or in an acute withdrawal state

   vi. Currently pregnant or planning to become pregnant.

   vii. Currently experiencing nicotine use disorder or any smoking of cigarettes or use of other nicotine containing products within a week before the eye tracking visit.

   viii. Has had ECT treatment within the last 6 months.
5. Inclusion and exclusion criteria for Group 5: Healthy Volunteers

   1. Inclusion criteria for Group 5:

   i. Male or female, age 18 or older

   ii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   iii. In the opinion of the investigator, has the competency to understand and sign the informed consent

   iv. Physically healthy as determined by research psychiatrist

   v. Without any current and/or lifetime psychiatric disorder as confirmed by the Mini International Neuropsychiatric Interview (MINI)

   b. Exclusion Criteria for Group 5:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Any psychiatric disorder including any severe personality disorder

   iv. Currently pregnant or planning to become pregnant

   v. Tests positive for illegal substances or prescription medications for which they do not have a valid prescription

   vi. Currently taking any steroids, stimulants, or opioid pain killers.

   vii. Currently experiencing nicotine use disorder or any smoking of cigarettes or use of other nicotine containing products within a week before the eye tracking visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects will those living in the greater Cleveland, OH area who respond to IRB approved advertising.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Measure the differences in attentional bias among the 5 groups by assessing how long it takes a subject to locate and fixate on each face on the screen | Baseline
  This paradigm involves the simultaneous presentation of 2 facial images. Two facial expressions (happy-neutral, sad-neutral, fearful-neutral, and neutral-neutral) from the same actor are presented simultaneously on each side of the screen. For each participant, happy, sad, fearful, and neutral facial expressions are randomly assigned to each side with each emotion category presented on each side with equal frequency. Each trial presents happy-neutral, sad-neutral, fearful-neutral and neutral-neutral facial expression in a new random order for each participant. Each trial begins with a central cross, followed by presentation of facial stimuli for 250-500 ms. Direction of gaze is measured with x and y coordinates. The latency and velocity of eye movement will be measured. Eye movements that are stable for more than 100 msec within 1˚of visual angle are classified as a fixation. The time to locate the face and fixation time to each face will be compared.
Measure the differences in reward sensitivity among the 5 groups by assessing the amplitude of the saccade to reward and non-reward stimuli | Baseline
  The reward paradigm is to measure amplitude and velocity of saccades toward reward stimuli. A saccade is a rapid eye movement made by the primate and human after they make their decision among several options. The participant will be told that he/she will be rewarded for a making a correct saccade in response to congruent conditional stimulus and she/he will not be rewarded for making a correct saccade in response to an incongruent stimulus. Each participant will have 5-10 trials to practice before the recording begins. The velocity and amplitude of saccade to reward and non-reward stimuli will be recorded for each trials. The mean velocity and amplitude to reward and non-reward stimuli among the different groups of patients will be compared.
Measure the differences in reward sensitivity among the 5 groups by assessing the velocity of the saccade to reward and non-reward stimuli | Baseline
  The reward paradigm is to measure amplitude and velocity of saccades toward reward stimuli. A saccade is a rapid eye movement made by the primate and human after they make their decision among several options. The participant will be told that he/she will be rewarded for a making a correct saccade in response to congruent conditional stimulus and she/he will not be rewarded for making a correct saccade in response to an incongruent stimulus. Each participant will have 5-10 trials to practice before the recording begins. The velocity and amplitude of saccade to reward and non-reward stimuli will be recorded for each trials. The mean velocity and amplitude to reward and non-reward stimuli among the different groups of patients will be compared.
Measure the differences in cognitive control among the 5 groups by assessing the amplitude of the antisaccade | Baseline
  Antisaccade (AS) performance is a sensitive marker for cognitive control of behavior and executive functioning. In contrast to saccade, antisaccade is an eye movement away from a target of reward or non-reward stimulus. Commonly used antisaccade paradigm includes cue, preparation, and response execution. In this protocol, the patients will learn to make an antisaccade to a reward or non-reward stimulus. Patients will receive a reward for each correct antisaccade movement to reward stimuli. The paradigm will include equal number of reward and non-reward trials. Trials are pseudorandomized across runs. For the reward condition, the value of any single correct response is intentionally ambiguous to prevent subjects from keeping a running total of earnings during the task.
Measure the differences in cognitive control among the 5 groups by assessing the velocity of the antisaccade | Baseline
  Antisaccade (AS) performance is a sensitive marker for cognitive control of behavior and executive functioning. In contrast to saccade, antisaccade is an eye movement away from a target of reward or non-reward stimulus. Commonly used antisaccade paradigm includes cue, preparation, and response execution. In this protocol, the patients will learn to make an antisaccade to a reward or non-reward stimulus. Patients will receive a reward for each correct antisaccade movement to reward stimuli. The paradigm will include equal number of reward and non-reward trials. Trials are pseudorandomized across runs. For the reward condition, the value of any single correct response is intentionally ambiguous to prevent subjects from keeping a running total of earnings during the task.

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center - Mood Disorders Program, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No